CLINICAL TRIAL: NCT03491124
Title: Battlefield Acupuncture for Low Back Pain
Acronym: BFA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Geneva Foundation (Other)
Collaborators: TriService Nursing Research Program (Other)
Responsible Party: Principal Investigator, David Wilson, Research Coordinator, The Geneva Foundation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N16-006
Record Dates: First submitted 2018-03-23; First posted 2018-04-09 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Low Back Pain; Chronic Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Acupuncture, Ear

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham Treatment (Sham Comparator): Participants will continue to receive usual care from their primary care provider, which can include medications, physical therapy, biofeedback, and education according to DoD/VA guidelines for LBP management. Participants randomized to this arm will also receive a sham intervention, pointing a laser pointer to the ear without turning the laser on.
  Interventions: Other: Sham Treatment
- Auricular Acupuncture (Experimental): Participants will continue to receive usual care from their primary care provider, which can include medications, physical therapy, biofeedback, and education according to DoD/VA guidelines for LBP management. Participants randomized to this arm will receive up to five ASP needles per ear placed in the predetermined BFA pattern. Needles are placed until the participant states pain is reduced 1/10.
  Interventions: Other: Auricular Acupuncture

INTERVENTIONS:
Other: Auricular Acupuncture — Up to five small ASP needles placed in each ear until pain is reduced to 1/10.
  Other Names: Battlefield Acupuncture (BFA)
  Arms: Auricular Acupuncture
Other: Sham Treatment — Laser pointer pointed at the ear, but not turned on.
  Arms: Sham Treatment

SUMMARY:
The purpose of this study is to determine the effect of Battlefield Acupuncture (BFA) on outcomes for pain, sleep, and physical activity level in an active duty military sample with subacute or chronic lower back pain (LBP). BFA is a form of auricular acupuncture (AA) that has been implemented in many Department of Defense (DoD)/Veterans Affairs (VA) medical settings to alleviate acute or chronic pain. BFA uses five predetermined locations in a defined sequence to place semi-permanent needles in the ear. Subacute lower back pain is pain that has persistently lasted from four to twelve weeks. Chronic lower back pain is pain that lasts more than 12 weeks.

Hypothesis 1: Participants with subacute or chronic LBP will have reduced pain using BFA as compared to placebo.

Hypothesis 2: Participants with subacute or chronic LBP will have improved physical activity using BFA as compared to placebo.

Hypothesis 3: Participants with subacute or chronic LBP will have improved sleep quality as compared to placebo.

The secondary study aims are:

1. To explore the effects of BFA two weeks following the treatment for LBP.

   1. Do positive outcomes appreciated with BFA persist over two weeks?
   2. What is the pain medication usage during and after intervention treatments?
2. To explore the effectiveness of BFA on trunk flexion mobility and balance.

   1. Does pain reduction improve trunk flexion and balance?
   2. Does improved truck flexion mobility and balance contribute to increased physical activity?

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of LBP (pain for > 4 weeks, with or without radiating nerve pain
* Age 18 to 50 years
* Active duty military, Public Health Service, or Coast Guard (guard and reserve on active orders)
* Pain score 3/10 or higher as patient reported on the DVPRS
* mODI score ≥ 20%
* No anticipated prolonged temporary duty, deployment, or vacation within the next month.

Exclusion Criteria:

* Any severe comorbidity
* LBP neurologic "red flags" indicating serious spinal pathology (i.e. bowel or bladder dysfunction)
* Auricular acupuncture in the past 6 months
* Use of steroids in the month prior to the study
* Hemorrhagic disorders
* Malignancy
* Unexplained weight loss
* Severe scoliosis or congenital spine disorder
* Back pain because of a visceral problem (e.g. endometriosis)
* Under surgeon's care for back surgery within the last 12 months
* Balance disorder
* Pregnancy or suspected pregnancy (last menstrual period will be reported by the patient)
* Aversion to needles
* Previous keloid scar formation
* Active infection on the ear
* Bleeding disorder
* Metal allergy
* Mental health diagnosis requiring medication (depression, PTSD, etc)
* Untreated sleep apnea or other sleep disorders

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2018-03-23 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Pain level change over time on the Defense/Veterans Pain Rating Scale(DVPRS). | The DVPRS will be administered weekly for seven times. Followed by a one time washout 2 weeks later.
  Participant reported pain level using the DVPRS. DVPRS pain level ranks from 0 (no pain) to 10 (As bad as it can be. Nothing else matters).

SECONDARY OUTCOMES:
Change in pain medication need. | A medication form will be administered weekly for seven times. Followed by a one time washout 2 weeks later.
  A self reported increase, decrease, or no change in medication use.
Change in trunk flexion. | Trunk flexion will be administered weekly for seven times. Followed by a one time washout 2 weeks later. If the participant has a DVPRS >=2 and mODI >=20%, trunk flexion will also be measured after the intervention.
  Trunk flexion will be assessed with Dual Digital Inclinometers. The Dual Digital Inclinometer is placed around the sacrum and measures the angle of flexion.
Change in balance | The FRT and TUG will be administered weekly for seven times. Followed by a one time washout 2 weeks later. If the participant has a DVPRS >=2 and mODI >=20%, the FRT and TUG will also be measured after the intervention.
  Balance is measured by Functional Reach Test(FRT) and Timed Up and Go Test(TUG). The FRT assesses a patient's stability by measuring the maximum distance an individual can reach forward while standing in a fixed position. The TUG is a simple test used to assess a person's mobility and requires both static and dynamic balance. It measures the time that a person takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down.
Change in physical activity | The mODI will be administered weekly for seven times. Followed by a one time washout 2 weeks later. The Actigraph watch is worn the entire 8 weeks.
  Activity will be measured using an Actigraph watch and Modified Oswestry Low Back Pain Disability Questionnairre(mODI)
Change in sleep quality | The ESS and ISI will be administered weekly for seven times. Followed by a one time washout 2 weeks later. The Actigraph watch is worn the entire 8 weeks.
  Sleep will be measured using an Actigraph watch, Epworth Sleepiness Scale(ESS), and Insomnia Severity Index(ISI)

OTHER OUTCOMES:
Health and well being | The SF-8 is administered the first, fourth, and eighth week.
  Health and well being is measured using the SF-8 Health Survey (4 Week Recall).
Height, weight, and Body Mass Index(BMI) | Height, weight, and BMI is measured the first and eighth week.
  The participants height and weight is measured. A BMI is also calculated using the following formula: BMI = kg/m2 where kg is a person's weight in kilograms and m2 is their height in meters squared.

CONTACTS AND LOCATIONS:
Overall Officials: Candy Wilson, PhD, Principal Investigator — Uniformed Services University of the Health Sciences
Locations (1):
- Malcolm Grow Medical Clinics and Surgery Center, Andrews Air Force Base, Maryland, United States